CLINICAL TRIAL: NCT06626646
Title: Vascular Regenerative Cell Exhaustion in Adults with Peripheral Artery Disease
Brief Title: Vascular Regenerative Cell Exhaustion in Adults with Peripheral Artery Disease (PAD-VRCE)
Acronym: PAD-VRCE
Status: Recruiting | Type: Observational
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00080564
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Vascular Diseases; Cardiovascular Disease; Type 2 Diabetes; Peripheral Artery Disease
Keywords: Progenitor cells; Cardiovascular disease; Peripheral artery disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Peripheral Artery Disease: 20 patients with clinically significant/symptomatic Peripheral Artery Disease defined as symptomatic claudication and an ABI of <0.85
- Control Group: 20 patients who do not have Peripheral Artery Disease

SUMMARY:
PAD-VRCE is an observational, cross-sectional, two arm study aimed at determining if the presence of peripheral artery disease (PAD) can influence the number of circulating regenerative cells in blood. From peripheral blood samples, circulating progenitor cell content will be assessed via flow cytometry and compared between individuals with PAD and individuals without PAD. Ultimately, this study plans to evaluate the relationship between PAD, vascular regenerative cell exhaustion and overall cardiovascular health.

DETAILED DESCRIPTION:
Individuals with peripheral artery disease (PAD) have been shown to have poorer cardiovascular health outcomes than the general population. It is believed that the number of people living with PAD is greatly underestimated and furthermore, mortality due to the most severe form of PAD - critical limb ischemia - is increasing. There is a growing body of evidence that the presence of cardiovascular risk factors leads to the imbalance of circulating regenerative cells. The aggregate impact of this regenerative cell exhaustion phenotype is an increased risk of adverse events and progression of disease states.

PAD-VRCE is an observational, cross-sectional, two-arm cohort study aimed at determining the differences in the progenitor cell profiles in the blood of individuals with PAD in comparison to individuals without PAD. We hypothesize that people with PAD will exhibit depleted levels of these progenitor cells defined as vascular regenerative cell exhaustion. VRCE impacts the function of anti-inflammatory cells and associated repair mechanisms within blood vessels, and may contribute to the differential long term outcomes between the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 and ≤80 years of age who meet either of the following criteria:

   1. Clinically significant/symptomatic PAD (defined as symptomatic claudication with and an ankle brachial index of less than 0.85).
   2. No history of PAD.
2. Willing and able to provide written informed consent and comply with study procedures.

Exclusion Criteria:

1. Unable or unwilling to provide written informed consent or to provide a peripheral blood sample.
2. Any life-threatening disease expected to result in death within two years.
3. Any malignancy not considered cured (except basal cell carcinoma of the skin). An individual is considered cured if there has been no evidence of cancer recurrence for the five years prior to screening.
4. Uncontrolled hypertension.
5. New York Heart Association Class IV heart failure.
6. Active liver disease or liver dysfunction.
7. Active kidney disease or kidney dysfunction.
8. History of hemorrhagic stroke or other major bleeding disorder.
9. White blood cell count of ≥15x10^9/L.
10. Active infectious disease requiring systemic antibiotic or anti-viral agents.
11. Known acquired immunodeficiency syndrome, such as Human Immunodeficiency Virus.
12. On oral steroid therapy (e.g. prednisone or other corticosteroids) or other immunosuppressive agents (e.g. methotrexate).
13. Treated autoimmune disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from primary care and cardiology outpatient clinics in the Greater Toronto Area using paper-based and electronic medical records.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The difference in the frequency / absolute number of circulating primitive myeloid progenitor cells (ALDHhiSSClow) between individuals with PAD and without PAD | Baseline

SECONDARY OUTCOMES:
The difference in the amount of intracellular reactive oxygen species produced by ALDHhi progenitor cell subsets in individuals with PAD and without PAD | Baseline
The difference in the levels of circulating inflammatory and oxidative stress markers in individuals with PAD and without PAD | Baseline
The difference in the frequency /absolute count of ALDHhiSSCmid monocytes in individuals with PAD or without PAD | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, Principal Investigator — University of Toronto; David A Hess, PhD, Principal Investigator — Western University, Canada
Locations (2):
- Canada (2):
  - North York Diagnostic and Cardiac Centre, North York, Ontario
  - Diagnostic Assessment Centre, Scarborough Village, Ontario

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krishnaraj A, Bakbak E, Teoh H, Pan Y, Firoz IN, Pandey AK, Terenzi DC, Verma R, Bari B, Bakbak AI, Kunjummar SP, Yanagawa B, Connelly KA, Mazer CD, Rotstein OD, Quan A, Bhatt DL, McGuire DK, Hess DA, Verma S. Vascular Regenerative Cell Deficiencies in South Asian Adults. J Am Coll Cardiol. 2024 Feb 20;83(7):755-769. doi: 10.1016/j.jacc.2023.12.012. PMID 38355246
- [Background] Hess DA, Terenzi DC, Trac JZ, Quan A, Mason T, Al-Omran M, Bhatt DL, Dhingra N, Rotstein OD, Leiter LA, Zinman B, Sabongui S, Yan AT, Teoh H, Mazer CD, Connelly KA, Verma S. SGLT2 Inhibition with Empagliflozin Increases Circulating Provascular Progenitor Cells in People with Type 2 Diabetes Mellitus. Cell Metab. 2019 Oct 1;30(4):609-613. doi: 10.1016/j.cmet.2019.08.015. Epub 2019 Aug 30. PMID 31477497
- [Background] Hicks CW, Yang C, Ndumele CE, Folsom AR, Heiss G, Black JH 3rd, Selvin E, Matsushita K. Associations of Obesity With Incident Hospitalization Related to Peripheral Artery Disease and Critical Limb Ischemia in the ARIC Study. J Am Heart Assoc. 2018 Aug 21;7(16):e008644. doi: 10.1161/JAHA.118.008644. PMID 30369315
- [Background] Shishehbor MH, White CJ, Gray BH, Menard MT, Lookstein R, Rosenfield K, Jaff MR. Critical Limb Ischemia: An Expert Statement. J Am Coll Cardiol. 2016 Nov 1;68(18):2002-2015. doi: 10.1016/j.jacc.2016.04.071. Epub 2016 Sep 28. PMID 27692726
- [Background] Fowkes FG, Rudan D, Rudan I, Aboyans V, Denenberg JO, McDermott MM, Norman PE, Sampson UK, Williams LJ, Mensah GA, Criqui MH. Comparison of global estimates of prevalence and risk factors for peripheral artery disease in 2000 and 2010: a systematic review and analysis. Lancet. 2013 Oct 19;382(9901):1329-40. doi: 10.1016/S0140-6736(13)61249-0. Epub 2013 Aug 1. PMID 23915883